CLINICAL TRIAL: NCT06875466
Title: Exploring the Health Benefits of Sauna Bathing - a Pilot Study
Brief Title: Exploring the Health Benefits of Sauna Bathing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Centre for Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Sauna
Record Dates: First submitted 2025-03-09; First posted 2025-03-13 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sauna Bathing (Experimental): Participants receive the sauna bathing treatment (1 session per week for 8 weeks)
  Interventions: Device: Sauna bathing

INTERVENTIONS:
Device: Sauna bathing — Finnish sauna bathing, participants will sauna once per week for 8 weeks

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of mortality in Aotearoa New Zealand, with hypertension being a major risk factor that remains difficult to manage with medication. Finnish sauna bathing (FSB), a widely practiced form of heat therapy, has been linked to lower risks of CVD, stroke, and overall mortality. Traditionally, FSB is combined with cold water immersion (CWI), but the combined effects of these therapies remain under explored. While sauna research often focuses on physiological aspects, this study aims to take a holistic approach to understanding its impact on cardiovascular health.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) remains the leading cause of mortality and morbidity in Aotearoa New Zealand. High blood pressure is a significant risk factor for CVD, with nearly half of older adults in Aotearoa diagnosed with hypertension, and it being relatively intractable to attempts thus far at treatment via antihypertensive medications.

Finnish sauna bathing (FSB) is one form of heat therapy, characterised by the use of a wood-fired sauna in which water is thrown over hot stones to create steam. In Finland, the sauna is not only a common therapy but also deeply ingrained in the cultural fabric, with many households having their own sauna. Traditionally, saunas were communal places where people came together to relax and share experiences thus fostering social connections. Lifelong sauna use is associated with markedly lower risk for chronic diseases such as; CVD, stroke, and all-cause mortality. Integral to the FSB experience is the practice of cold water immersion (CWI) which typically involves a plunge into icy waters, or exposure to freezing temperatures, in between sauna bathing.

Sauna bathing is typically researched with a physiological / biomedical lens and in isolation, that is, the additive effects of sauna bathing and cold-induced adaptations from cold-water immersion are not well understood, highlighting a gap in this research area. Additionally, the health benefits of sauna are wide ranging, therefore our focus is to use a holistic lens to explore the impact of sauna bathing cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

* SBP: 110-179 mmHg; DBP 60-99 mmHg)
* 18 - 70 y old.
* Participants who are prescribed anti-hypertensive or dyslipidaemia medications will be included but must be on a stable dose for at least 30 days.

Exclusion Criteria:

* stable or unstable angina
* recent myocardial infarction (<3 months)
* orthostatic hypotension
* severe aortic stenosis
* pregnancy
* acute infectious diseases
* rheumatoid arthritis in the acute inflammatory phase
* fever for any reason
* any other medical condition deemed a risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
24 hour ambulatory blood pressure | 8 weeks
  This measure will be taken before and after the intervention. There are four sections of the questionnaire. The first two sections use the scale 1 - 5 where 1 = never, 2 = rarely, 3 = occasionally, 4 = regularly, 5 = constantly. A higher score means a worse outcome. Section three uses the scale 1 - 5 where 1 = not at all, 2 = not really, 3 = sometimes, 4 = yes, 5 = yes, absolutely; in this section a higher score means a better outcome. Section four uses a scale 1 - 5 where 1 = strongly disagree, 2 = disagree, 3 = not sure, 4 = agree, 5 = strongly agree; a higher score means a better outcome.

SECONDARY OUTCOMES:
Quality of life questionnaire | 8 weeks
  This measure will be taken before and after the intervention
PROMIS Sleep Questionnaire | 8 weeks
  This measure will be taken before and after the intervention. There are four questions which uses the scale is from 1 -5. 1 = Not at all, 2 = a little bit, 3 = somewhat, 4 = quite a bit, 5 = very much. There are three questions that use the scale 1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5 = always. One questions uses the scale 1 = very poor, 2 = poor, 3 = fair, 4 = good, 5 = very good. In all questions the higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Rolleston, PhD, Principal Investigator — The Centre for Health
Locations (1):
- The Centre for Health, Tauranga, New Zealand

IPD SHARING:
Plan to Share IPD: No